CLINICAL TRIAL: NCT06969066
Title: Effect of Cognitive Remediation Therapy (CRT) for Chronic Insomnia (CI) With Cognitive Impairment
Brief Title: Memory Training in Insomnia With Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-CRT
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Therapy/Methods; Insomnia Chronic; Cognitive Dysfunction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT plus Sleep Hygiene Education (Experimental)
  Interventions: Behavioral: Cognitive Remediation Therapy plus Sleep Hygiene Education (CRT+SHE)
- Sleep Hygiene Education Only (Active Comparator)
  Interventions: Behavioral: Sleep Hygiene Education Only (SHE)

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy plus Sleep Hygiene Education (CRT+SHE) — Participants will receive Cognitive Remediation Therapy (CRT) combined with Sleep Hygiene Education (SHE). CRT includes structured training sessions targeting attention, memory, visuospatial skills, calculation ability, logical reasoning, and language abilities. Sessions will be conducted daily for 50 minutes over 6 weeks. Sleep Hygiene Education will cover standard recommendations to improve sleep behaviors.
  Arms: CRT plus Sleep Hygiene Education
Behavioral: Sleep Hygiene Education Only (SHE) — Participants will receive Sleep Hygiene Education (SHE) only, including guidance on adjusting sleep schedules, maintaining healthy sleep environments, minimizing stimulant intake, and managing sleep-related behaviors, without any CRT intervention.
  Arms: Sleep Hygiene Education Only

SUMMARY:
This randomized controlled trial investigates the effects of Cognitive Remediation Therapy (CRT) on chronic insomnia (CI) with mild cognitive impairment.

DETAILED DESCRIPTION:
Chronic insomnia (CI) is a prevalent sleep disorder that not only causes night-time sleep difficulties but also impairs daytime functioning and cognitive abilities, including deficits in attention, memory, and executive function. Persistent insomnia may diminish the brain's information processing capacity, affecting memory, attention, and decision-making. CRT, a structured cognitive training intervention, has been shown in psychiatric populations to enhance memory, attention, and executive function by promoting neuroplasticity, neurotransmitter modulation, and optimizing brain activity patterns.

Applying CRT to CI patients may similarly support cognitive recovery and indirectly improve sleep quality. However, empirical evidence remains limited.

This randomized controlled trial will enroll 70 patients with CI and cognitive decline. Participants will be randomly assigned to either a CRT plus Sleep Hygiene Education (SHE) group or an SHE-only group (n=35 each). The CRT intervention will last 6 weeks, with daily 50-minute sessions. Evaluations will occur at baseline, post-intervention, and at 3, 6, and 12 months follow-up. This study aims to provide evidence for CRT as a treatment for CI with cognitive impairment and inform future clinical practices.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for Insomnia Disorder according to DSM-5.
2. Pittsburgh Sleep Quality Index (PSQI) total score > 5.
3. Age ≥ 8 years.
4. Voluntary participation with signed informed consent.
5. Meets the cognitive impairment criteria associated with CI:

(1) Right-handedness. (2) Age between 55 and 75 years. (3) Education duration ≥ 12 years. (4) At least junior high school education level; fulfills Petersen's diagnostic criteria for mild cognitive impairment: 1.Subjective complaints of memory decline. 2.Duration of cognitive complaints ≥ 3 months. 3.Assessment scores: Global Deterioration Scale (GDS) rating of stage 1-2; Clinical Dementia Rating (CDR) score of 0-0.5. 4.Memory test scores falling ≥ 1.5 standard deviations below the age- and education-matched norms: MMSE ≥ 24, MoCA < 26, Activities of Daily Living (ADL) score > 26. 5.Memory impairment as the primary deficit, with relatively preserved functioning in other cognitive domains.

6.Normal daily functional abilities. 7.Exclusion of dementia or any major physical or psychiatric disorders that could impair brain function.

Exclusion Criteria:

1. Presence of severe physical illnesses or major psychiatric disorders, or assessed risk of suicide.
2. Diagnosed or suspected sleep breathing disorders, restless legs syndrome, circadian rhythm sleep disorders, or currently engaged in shift work.
3. Pregnancy or breastfeeding.
4. Currently undergoing any form of psychological therapy.
5. History of infectious diseases such as syphilis or HIV.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The change of Pittsburgh Sleep Quality Index (PSQI) total scores from baseline to 6 weeks. | Baseline, 6 weeks
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.

SECONDARY OUTCOMES:
The change of PSQI total scores from baseline to 3 months, 6 months, and 12 months. | Baseline, 3 months, 6 months, 12 months
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.
The change of Insomnia severity index (ISI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The ISI reporting insomnia symptoms severity consists of 7-items on a 5-point Likert scale, and the total score ranges from 0 to 28 with higher scores indicating more severe insomnia.
The change of sleep efficiency from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
The change of Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The DBAS assessing sleep related cognitions in 16 items rated on a 10-point Likert scale, and the total score ranges from 0 to 160 with higher scores indicating more intensive dysfunctional beliefs.
The change of Snaith-Hamilton Pleasure Scale (SHAPS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The SHAPS assessing anhedonia consists of 14 items, and the total score ranges from 14 to 56 with higher scores indicating more serious the anhedonia.
The change of Short Form 36 (SF-36) total scores from baseline to 6 weeks, 3 months, 6 months, 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months.
  The SF-36 quantifying the quality of life in relation to health status consists of 36-items with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The total score ranges from 0-100 (the worst possible to the most possible).
The change of Patient Health Questionnaire-4 (PHQ-4) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-4 comprises a 2-item depression scale and a 2-item anxiety scale. Each instrument can reach values from 0-6. Higher Scores are indicating higher distress.
The change of Beck Depression Inventory (BDI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BDI assessing the existence and severity of symptoms of depression consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe depressive symptoms.
The change of Beck Anxiety Inventory (BAI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BAI assessing the existence and severity of symptoms of anxiety consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe anxiety.
The change of Patient Health Questionnaire-15 (PHQ-15) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-15 measuring somatic distress consists of 15 items, and the total score ranges from 0 to 30 with higher scores indicating more severe somatic distress.
The change of 5-item Perceived Deficits Questionnaire-Depression (PDQ-D-5) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PDQ-D-5 assessing perceived cognitive deficits from the patient's perspective consists of 5 items, and the total score ranges from 0 to 20 with higher scores indicating greater perceived deficit.
The change of Life Events Scale (LES) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The LES assessing the perceived stress and number of stressful life events experienced consists of 48 items which are classified into three dimensions: family life events (28 items), work and study events (13 items), and social events (7 items) with higher scores in LES perceived greater stressfulness

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No